CLINICAL TRIAL: NCT04434222
Title: Effect of Compliance Controlled Postoperative Compressive Stockings Therapy After Total Knee Arthroplasty: a Randomized Controlled Trial
Brief Title: Compressive Stockings Therapy After TKA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough study participants and missing compliance to perform analysis
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W759
Record Dates: First submitted 2020-04-28; First posted 2020-06-16 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Compliance of Wearing of Compressive Stockings; Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compressive stockings group (Active Comparator): Group receives postoperatively compressive stockings for a period of 6 weeks.
  Interventions: Device: Compressive stockings
- Control group (No Intervention): The control group is treated without compressive stockings.

INTERVENTIONS:
Device: Compressive stockings — Compressive stockings with built in Orthotimer Sensor
  Arms: Compressive stockings group

SUMMARY:
Due to swelling after total knee arthroplasty, postoperative mobilization and training is impeded in addition to higher pain level in patients. With postoperative compressive stockings to prevent oedema, haematoma and postoperative pain we would like to investigate if compressive stockings reduce postoperative swelling and pain and furthermore improve mobilization and knee function.

In this randomized controlled trial, 88 patients are randomized in two groups. One group receives postoperatively compressive stockings for a period of 6 weeks. The control group is treated without compressive stockings. The patients compressive stockings wearing compliance is controlled with a temperature sensitive sensor. The patients will be informed about the implantation of the sensor.

Outcome measures are knee- calf- and ankle swelling in mm, pain, WOMAC and KSS score preoperatively and at 12 weeks, 12 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a total knee replacement
* Written consent of the study participant

Exclusion Criteria:

* Peripheral arterial disease II, III or IV
* Diabetes mellitus
* Systemic inflammatory diseases
* Benign or malignant neoplasms
* Revision interventions
* Right heart failure
* pulmonary edema
* Open / chronic skin lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Knee Function KSS 6 weeks postoperative | 6 weeks postoperative
  Knee Society Score - KSS
Knee Function KSS 12 weeks postoperative | 12 weeks postoperative
  Knee Society Score - KSS
Knee Function KSS 1 year postoperative | 1 year postoperative
  Knee Society Score - KSS
Knee Function WOMAC 6 weeks postoperative | 6 weeks postoperative
  Western Ontario and McMaster Universities Osteoarthritis Index - WOMAC
Knee Function WOMAC 12 weeks postoperative | 12 weeks postoperative
  Western Ontario and McMaster Universities Osteoarthritis Index - WOMAC
Knee Function WOMAC 1 year postoperative | 1 year postoperative
  Western Ontario and McMaster Universities Osteoarthritis Index - WOMAC
Pain 6 weeks postoperative | 6 weeks postoperative
  Visuelle Analogskala - VAS (1-10)
Pain 12 weeks postoperative | 12 weeks postoperative
  Visuelle Analogskala - VAS (1-10)
Pain 1 year postoperative | 1 year postoperative
  Visuelle Analogskala - VAS (1-10)

SECONDARY OUTCOMES:
Swelling 6 weeks postoperative | 6 weeks postoperative
  Swelling in mm
Swelling 12 weeks postoperative | 12 weeks postoperative
  Swelling in mm
Swelling 1 year postoperative | 1 year postoperative
  Swelling in mm
Compliance first 6 weeks postoperativ | First 6 weeks postoperativ
  Measured with Orthotimer sensor

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik Balgrist, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No